CLINICAL TRIAL: NCT06123208
Title: The Influence of the Resistant Starch and Protein Content of Pulses on Substrate Oxidation
Brief Title: Impact of Eating Beans on Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GFHNRC513
Record Dates: First submitted 2023-10-30; First posted 2023-11-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole cooked pinto bean meal (Experimental): Participants will consume a meal comprised of 100 grams of whole cooked pinto beans
  Interventions: Other: Whole cooked pinto bean
- Pinto bean flour meal (Experimental): Participants will consume a meal comprised of pinto bean flour equivalent to 100 grams of whole cooked pinto beans
  Interventions: Other: Pinto bean flour
- Control meal (Active Comparator): Participants will consume a control meal
  Interventions: Other: Control

INTERVENTIONS:
Other: Whole cooked pinto bean — Meal comprised of whole cooked pinto beans
  Arms: Whole cooked pinto bean meal
Other: Pinto bean flour — Meal comprised of pinto bean flour
  Arms: Pinto bean flour meal
Other: Control — Control meal
  Arms: Control meal

SUMMARY:
The purpose of this research is to test how eating a meal containing beans impacts how participants' bodies use food for energy.

DETAILED DESCRIPTION:
The objective of this project is to test whether consuming a whole food that naturally contains resistant starch (RS), such as pulses, increases fat oxidation. The primary hypothesis is that consuming a RS-rich meal in which the RS is derived from a whole food (i.e., pinto beans, pinto bean flour) will increase postprandial fat oxidation to a greater extent than consuming a meal low in RS but containing the same amount of energy and macronutrient content.

ELIGIBILITY:
Inclusion Criteria:

* BMI >18.5 or <30 kg/m2
* Ability to understand and sign the consent form
* Ability of transportation (i.e., participants must be able to provide their own transportation to the Grand Forks Human Nutrition Research Center)
* Non-smoking or use of other tobacco products, including e-cigarettes
* Not taking steroid-based medications; not planning to or currently attempting to gain or lose weight
* All females of childbearing age must be on birth control for a minimum of 3 months prior to start of study

Exclusion Criteria:

* Inability or unwillingness to consume any food item in the test meals
* More than a 10% change in body weight within the past 2 months
* Participation in a weight loss diet/exercise program
* Current or planned pregnancy
* Lactation
* Uncontrolled hypertension (systolic >160 mmHg or diastolic >100 mmHg)
* Diagnosed cardiovascular, pulmonary, skeletal and metabolic diseases
* Fasting glucose > 100 mg/dL or non-fasting (1-2 hours after eating) >140 mg/dL
* Using medications known to affect appetite, blood lipids, body composition, body weight, or food intake (appetite control drugs, steroids, antidepressants)
* Non-English speaking

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Acute effects of consuming processed pulse-based food products on substrate utilization | 5 hours after meal consumption
  The effect of consuming whole beans or bean-derived flour on the use of fat, carbohydrate, and protein for energy will be determine using whole room calorimetry. Fat, carbohydrate, and protein oxidation will be calculated as an absolute amount of grams per day and as a percentage of energy expenditure.

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT06123208/ICF_000.pdf